CLINICAL TRIAL: NCT01702220
Title: Calmer Life: A Randomized Controlled Trial of a Participant-Centered Treatment for Anxiety in Low-Income, Older Adults
Brief Title: Calmer Life: Testing the Effectiveness of a Treatment for Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Retirement Research Foundation (Other); Archstone Foundation (Other)
Responsible Party: Principal Investigator, Melinda Stanley, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H30928
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Generalized Anxiety Disorder; Anxiety Disorder NOS
Keywords: Generalized Anxiety Disorder; Geriatric
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Experimental)
  Interventions: Behavioral: CBT
- Enhanced Community Care (ECC) (Active Comparator)
  Interventions: Other: ECC

INTERVENTIONS:
Behavioral: CBT — 6-12 sessions of CBT in person or over the phone
  Other Names: Cognitive Behavior Treatment, Cognitive Behavior Therapy
  Arms: CBT
Other: ECC — 6 biweekly sessions of ECC over the telephone
  Other Names: Enhanced Community Care
  Arms: Enhanced Community Care (ECC)

SUMMARY:
The overall goals of the proposed research study are to: (1) examine quantitative outcomes in a well-conducted randomized clinical trial of Calmer Life, relative to Enhanced Community Care, an information and referral intervention that represents care in a real-world community-service environment, and (2) evaluate implementation feasibility, which includes training community providers; examining program reach, engagement, acceptability, and barriers-facilitators; and preparing practical tools for replicating the program.

DETAILED DESCRIPTION:
Cognitive behavioral treatment (CBT) produces positive outcomes for late-life worry/GAD in academic and primary care settings, but minorities are significantly underrepresented in clinical trials, and standard CBT poorly addresses the needs of low-income minority older adults in underserved communities. More attention needs to be given to service delivery of anxiety treatments for underserved older adults. Calmer Life (CL) is a culturally tailored, participant-centered research study that offers a skills-based intervention for late-life anxiety and includes other elements of care to meet the needs of underserved, minority older adults, including the option to integrate religion/spirituality (R/S), flexible delivery modes, and modular treatment format.

Participants will be randomly assigned to CL or Enhanced Community Care(ECC). CL and ECC will be provided by behavioral health clinicians recruited from partner organizations, psychology trainees, and other research staff over 3 months. Assessments will occur at baseline and 3 months.

Participants in the CL condition can choose up to 12 individual skill sessions, and will be recommended to complete a minimum of 6 sessions. If participants desire to incorporate R/S, an R/S assessment occurs during session 2 to help the provider understand the participant's beliefs and practices. R/S can be integrated into any of the skills learned during the intervention (e.g., deep breathing, self-statements, sleep management) or omitted entirely.

Participants in the ECC condition will receive brief biweekly check in calls to provide information about community resources (including mental health), offer emotional support, and assess symptom severity and need for crisis intervention. Emergency procedures will be followed in crisis situations. After 3 months of ECC is completed, participants in the ECC group will be offered the CL intervention.

Outcome measures will be administered for participants in both groups at baseline, 1 month, and 3 months. Participants in ECC will complete measures at 6 months after completion of CL.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older
* Principal or Co-principal diagnosis of GAD or ADNOS
* Must speak English
* Must have a health care or social service provider and provide written authorization to research team to communicate with their health-care or social service provider
* Must live, work, worship, attend community functions, and/or receive health care in target geographic areas

Exclusion Criteria:

* Active suicidal intent
* Current psychosis
* Mania or substance abuse within the last month
* Cognitive impairment according to a Mini Cog screener score of 3 or lower

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Geriatric Anxiety Inventory | 3 months
Penn State Worry Questionnaire (PSWQ-A) | 3 months
Generalized Anxiety Disorder-7 | 3 months

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | 3 months
Insomnia Severity Index | 3 months
Late-Life Functional Disability Index | 3 months
SF-12 Health Survey | 3 months
Client Satisfaction Questionnaire | 3 months
Brief RCOPE | 3 months
  Religious coping
Health services use | 3 months
Use of psychotropic medication | 3 months
Brief Multidimensional Measure of Religiousness and Spirituality | 3 months
Satisfaction with Life Scale | 3 months
Geriatric Depression Scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Melinda A Stanley, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Center for Quality of Care and Utilization Studies, Houston, Texas, United States

REFERENCES:
- [Derived] Stanley MA, Wilson N, Shrestha S, Amspoker AB, Armento M, Cummings JP, Evans-Hudnall G, Wagener P, Kunik ME. Calmer Life: A Culturally Tailored Intervention for Anxiety in Underserved Older Adults. Am J Geriatr Psychiatry. 2016 Aug;24(8):648-658. doi: 10.1016/j.jagp.2016.03.008. Epub 2016 Mar 29. PMID 27426212